CLINICAL TRIAL: NCT04568369
Title: Functional Near Infrared Spectroscopy as a Biomarker of Response in Patients With Post-concussion Syndrome Treated With Transcranial Magnetic Stimulation
Brief Title: Treatment of Post-concussion Syndrome With TMS: Using FNIRS as a Biomarker of Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-1552
Record Dates: First submitted 2020-09-04; First posted 2020-09-29 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Transcranial Magnetic Stimulation; Functional Near-Infrared Spectroscopy; Post-Concussion Syndrome; Concussion; Mild Traumatic Brain Injury; Post-traumatic Stress Disorder
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This study will be a double-blind, sham-controlled, concealed allocation, randomized, cross over clinical trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be randomized with a random number generator to receive either sham or rTMS. The research assistant administering the fNIRS and PTSD assessments, will be blinded to the treatment allocations. Once the study is completed, patients and all study personnel will be unblinded. Subjects in the sham group will be given the opportunity to cross over to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients will engage in a four-week treatment protocol (20 treatments). This was chosen as it is the midpoint between typical depression and migraine protocol durations. A standardized atlas brain with Montreal neurologic institute (MNI) coordinates will be used for navigation. The DLPFC will be located through MNI coordinates (-50, 30, 36). The intensity of the rTMS will be 100-120% of resting motor threshold amplitude, with a frequency of 10 Hz, 10 trains of 60 pulses/train (total of 600 pulses) and an inter-train interval of 45s.
  Interventions: Device: rTMS
- Sham group (Sham Comparator): In the sham condition, a sham coil will be applied to the scalp after the resting motor threshold is determined. Patients will be able to hear the sound and feel the vibration of sham coil, but will not experience any effective stimulation. Previous sham studies have demonstrated efficacy of the blinding method.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — See treatment arm description.

SUMMARY:
Every year, approximately 2 million people in the United States and 280,000 in Canada experience a mild traumatic brain injury/concussion. In patients with concussion, symptoms experienced following injury usually get better within 3 months. However, approximately 5-25% of people will experience symptoms beyond the 3 month period, characterized by persistent headaches, fatigue, insomnia, anxiety, depression, and thinking or concentration problems, which contribute to significant functional impairment. Chronic headache is the most common symptom following concussions. They can last beyond 5 years following injury, significantly impacting daily activities. To date, post-concussion symptoms have no known "cure".

One potential approach to treating post-concussion symptoms may involve using drug-free interventions, such as neuromodulation therapy. This has the goal of restoring normal brain activity. Repetitive transcranial magnetic stimulation (rTMS) is one method currently being explored as a treatment option. TMS is a procedure where brain electrical activity is influenced by a magnetic field. Numerous studies using rTMS to treat other disorders, such as dementia, stroke, cerebral palsy, addictions, depression and anxiety, have shown much promise. The primary objective of this study is to determine whether rTMS treatment can significantly improve persistent post-concussion symptoms. A secondary objective is to explore the relationship between potential changes in brain function and clinical markers associated with rTMS treatment and how functional near-infrared spectroscopy (fNIRS), a neuroimaging technology, may be used to assess rTMS-treatment response.

DETAILED DESCRIPTION:
Annually, up to 280,000 people in Canada and 42 million worldwide experience a mild traumatic brain injury (mTBI). In patients with mTBI, symptoms experienced following injury usually resolve within 3 months. However, up to 25% of patients will experience persistent post-concussion symptoms (PPCS), which can continue up to 1 year following injury. Common symptoms include headaches, dizziness, fatigue, irritability, depression, anxiety, emotional lability, concentration or memory difficulties, insomnia, and reduced alcohol tolerance (ICD-10 post-concussion syndrome diagnostic criteria). To date, there is no "cure" for PPCS and current treatment entails trial and error with behavior management, environmental modifications and medications. Consequently, there is a significant need for new approaches to symptom management in order to help improve functional impairment and disease burden, associated with PPCS. Transcranial magnetic stimulation (TMS) has been studied as an intervention for many mental health and neurological conditions, including major depression and migraines, and has shown initial promise for PPCS. We intend to study the efficacy of TMS for PPCS further in a randomized sham-controlled trial.

Mild traumatic injury is considered a risk factor in the development of post-traumatic stress disorder. As such, post-traumatic stress disorder and mild traumatic brain injury often co-occur and share similar symptoms, such as irritability, post-traumatic amnesia, sleep disturbances, concentration difficulties and cognitive processing deficits. Several studies have suggested the efficacy and safety of rTMS for the treatment of PTSD; however, a gap in the literature exists regarding treating comorbid post-traumatic stress disorder and PPCS following mild traumatic brain injury. To study potential differences in response to treatment between individuals experiencing PPCS with or without co-morbid post-traumatic stress disorder, we intend to measure PTSD symptoms for those with a clinical diagnosis of post-traumatic stress disorder. Tracking PTSD symptoms will allow insight into whether the presence of PTSD symptoms affects rTMS treatment outcomes in individuals experiencing PPCS.

RESEARCH QUESTIONS AND OBJECTIVES

The overall goal is to study the application of rTMS treatment to the left dorsal lateral prefrontal cortex (DLPFC) in patients with PPCS to improve overall symptom burden and to explore biomarkers of response, specifically functional near infrared spectroscopy (fNIRS).

Specifically the objectives are:

1. Primary Objective: to determine changes in brain physiology associated with rTMS treatment as recorded by fNIRS.
2. Secondary Objective: to determine whether patients with PPCS have significant improvement to a 20-day high frequency rTMS treatment protocol of the left DLPFC compared to patients with PPCS receiving a sham rTMS protocol as measured by the Rivermead post-concussion symptom questionnaire at 1 and 3 months post-treatment.
3. Third Objective: To determine what exploratory outcomes such as quality of life, headaches, anxiety, depression, sleep, and somatic symptoms also improve with TMS treatment in individuals suffering with PPCS. Quality of life will be measured via the Quality of Life after Brain Injury questionnaire (QOLIBRI), headache intensity will be measured via the Headache intensity Test - 6 (HIT-6), feelings of depression will be measured via the Patient Health Questionnaire -9 (PHQ-9), anxiety via the Generalized Anxiety Disorder -7 (GAD-7), sleep via the Sleep and Concussion Questionnaire and somatic symptoms which are commonly present in functional neurological disorders via the SOMS-CD and Patient Health Questionnaire-15 (PHQ-15). Since Functional Neurological Disorder is often associated with past trauma, trauma history will be assessed via the Brief Trauma Questionnaire (BTQ) and the Life Stress Questionnaire (LSQ).
4. To determine whether those with PPCS and PTSD respond differently to rTMS and what effect this has on their PTSD symptoms measured via the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) and the Montgomery-Asberg Depression Rating Scale. Participants with PTSD will be identified as those with scores higher than 33 in the PCL-5 and a clinical diagnosis of PTSD by a medical professional.
5. To examine potential blood biomarkers of post-concussion syndrome and post-traumatic stress disorder.

METHODS

This study will be a double-blind, sham-controlled, concealed allocation, randomized clinical trial.

Clinical Assessments: Demographic information will be collected prior to starting the study including age, sex, education, headache history, concussion history, past medical history, medication use, and family medical history. Baseline questionnaires will be completed including Headache Impact Test - 6 (HIT-6), Rivermead PPCS questionnaire, British Columbia post-concussion symptom inventory (BC-PSI), quality of life after brain injury questionnaire (QOLIBRI), patient health questionnaire-9 (PHQ-9), generalized anxiety disorder scale-7 (GADS-7),the St. Louis University Mental examination Tool (SLUMS), the screening for somatoform symptoms questionnaire (SOMS-CD), the post traumatic stress disorder checklist for DSM-5 (PCL-5), the Brief Trauma Questionniare (BTQ), the Life Stress Questionnaire (LSQ), the Patient Health Questionnaire-15 (PHQ-15), and the Sleep and Concussion Questionnaire (SCQ). Those who are identified as having a PCL-5 score of greater than 33, in addition to a clinical diagnosis of post-traumatic stress disorder, will also complete the LEC-5, CAPS-5, MADRS and Columbia Suicide Severity Rating Scale. Patients will be reassessed at the completion of their rTMS treatment, and at 1 and 3 months post-treatment. The questionnaires that will be completed at all follow-up visits include the Rivermead PPCS questionnaire, the HIT-6, the BC-PSI, the QOLIBRI, the PHQ-9, the GAD-7, the PCL-5, the SLUMS, the SOMS-CD, the PHQ-15, and the Sleep and Concussion Questionnaire. For the Sleep and Concussion Questionnaire, the initial screening section will not be completed at follow-ups. Participants in the PTSD sub-group will also complete the MADRS, CAPS-5 and Columbia Suicide Severity Rating Scale at the 1 month and 3-month follow-up visits.

TMS Protocol: Patients will engage in a four-week treatment protocol (20 treatments). This was chosen as it is the midpoint between typical depression and migraine protocol durations. A standardized atlas brain with Montreal Neurologic Institute (MNI) coordinates will be used for navigation. The DLPFC will be located through MNI coordinates (-50, 30, 36). The intensity of the rTMS will be 100-120% of resting motor threshold amplitude, with a frequency of 10 Hz, 10 trains of 60 pulses/train (total of 600 pulses) and inter-train interval of 45s. In the sham condition, a sham coil will be applied to the scalp after the resting motor threshold is determined. Patients will be able to hear the sound and feel the vibration of sham coil, but will not experience any effective stimulation. Previous sham studies have demonstrated efficacy of the blinding method.

Imaging: Functional near infrared spectroscopy (fNIRS) measurements will be recorded at baseline, immediately following rTMS, and at one month and 3-month follow-ups post-rTMS to investigate changes in brain physiology associated with rTMS treatment. fNIRS data will be recorded over the frontoparietal cortex at a sampling rate of 3.91 Hz, using the TechEn fNIRS system (TechEn Inc., Milford, MA USA). Each recording will consist of a 5 min rest period, followed by a finger tapping exercise, and a graded working memory task, previously described by Hocke et al (2018). The fNIRS data will be processed and analyzed for task-evoked activation using an ordinary least squares method of general linear modeling, as implemented in the NIRS Brain AnalyzIR Toolbox.

Blood Samples: Blood samples will be collected from a certified phlebotomist at the Heritage Medical Research Clinic located in the Cal Wenzel Precision Health building at the Foothills Medical Centre Campus. Analysis will focus on blood biomarkers of inflammation and CNS injury.

Statistical Analysis: Outcome parameters within each specific group (rTMS, sham, sex, PTSD diagnosis) will be analyzed by a one-way repeated measures analysis of variance (RM-ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of persistent post-concussion syndrome based on the ICD-10 criteria. This diagnosis should be given to the patient from a clinical practitioner.
* Concussion in the past 5 years attributed to current symptoms.
* Age 18-75 yrs.
* Current pharmacologic management can remain stable throughout the protocol such as use of abortive headache medications (i.e. triptans, opioids, tricyclic antidepressants, anti-seizure medications).

Exclusion Criteria:

* Prior history of TMS therapy
* TMS-related contraindications (pacemaker, metallic implant)
* Other medical conditions such as structural brain disease, previous seizures, psychiatric disorders excluding depression, PTSD and anxiety (schizophrenia, bipolar disorder), liver or kidney disease, malignancy, uncontrolled hypertension or diabetes, and pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Rivermead Post-Concussion Symptom Questionnaire (RPQ) | Baseline
  Assesses the severity of 16 commonly experienced PCS symptoms. Participants are instructed to rate the extent to which they have suffered from each of the listed symptoms in the past 24 hours, as compared to pre-injury levels, using a scale of 0 ("not experienced at all") to 4 ("a severe problem"). The RPQ has been demonstrated as a valid measure of PPCS with a minimal clinically important difference (MCID) of 4.5 points. It is advised to analyze this assessment as two separate scales (RPQ-13 and RRQ-3). The RPQ-3 has a total possible score of 0-12, with higher scores indicative of worse outcomes. The RPQ-13 has a total possible score of 0-52, with higher scores indicative of worse outcomes. Using these sub-scales, the instrument has good test-retest reliability and external construct validity. This questionnaire probes the separate cognitive, emotional and somatic components of PPCS.
Rivermead Post-Concussion Symptom Questionnaire (RPQ) | Within 1 week post-intervention
  Assesses the severity of 16 commonly experienced PCS symptoms. Participants are instructed to rate the extent to which they have suffered from each of the listed symptoms in the past 24 hours, as compared to pre-injury levels, using a scale of 0 ("not experienced at all") to 4 ("a severe problem"). The RPQ has been demonstrated as a valid measure of PPCS with a minimal clinically important difference (MCID) of 4.5 points. It is advised to analyze this assessment as two separate scales (RPQ-13 and RRQ-3). The RPQ-3 has a total possible score of 0-12, with higher scores indicative of worse outcomes. The RPQ-13 has a total possible score of 0-52, with higher scores indicative of worse outcomes. Using these sub-scales, the instrument has good test-retest reliability and external construct validity. This questionnaire probes the separate cognitive, emotional and somatic components of PPCS.
Rivermead Post-Concussion Symptom Questionnaire (RPQ) | 1-month post-intervention
  Assesses the severity of 16 commonly experienced PCS symptoms. Participants are instructed to rate the extent to which they have suffered from each of the listed symptoms in the past 24 hours, as compared to pre-injury levels, using a scale of 0 ("not experienced at all") to 4 ("a severe problem"). The RPQ has been demonstrated as a valid measure of PPCS with a minimal clinically important difference (MCID) of 4.5 points. It is advised to analyze this assessment as two separate scales (RPQ-13 and RRQ-3). The RPQ-3 has a total possible score of 0-12, with higher scores indicative of worse outcomes. The RPQ-13 has a total possible score of 0-52, with higher scores indicative of worse outcomes. Using these sub-scales, the instrument has good test-retest reliability and external construct validity. This questionnaire probes the separate cognitive, emotional and somatic components of PPCS.
Rivermead Post-Concussion Symptom Questionnaire (RPQ) | 3-months post-intervention
  Assesses the severity of 16 commonly experienced PCS symptoms. Participants are instructed to rate the extent to which they have suffered from each of the listed symptoms in the past 24 hours, as compared to pre-injury levels, using a scale of 0 ("not experienced at all") to 4 ("a severe problem"). The RPQ has been demonstrated as a valid measure of PPCS with a minimal clinically important difference (MCID) of 4.5 points. It is advised to analyze this assessment as two separate scales (RPQ-13 and RRQ-3). The RPQ-3 has a total possible score of 0-12, with higher scores indicative of worse outcomes. The RPQ-13 has a total possible score of 0-52, with higher scores indicative of worse outcomes. Using these sub-scales, the instrument has good test-retest reliability and external construct validity. This questionnaire probes the separate cognitive, emotional and somatic components of PPCS.

SECONDARY OUTCOMES:
Quality of Life After Brain Injury (QOLIBRI) | Baseline
  Assesses quality of life. Total possible score ranges between 0-100, with higher scores indicative of better outcomes.
Quality of Life After Brain Injury (QOLIBRI) | Within 1 week post-intervention
  Assesses quality of life. Total possible score ranges between 0-100, with higher scores indicative of better outcomes.
Quality of Life After Brain Injury (QOLIBRI) | 1-month post-intervention
  Assesses quality of life. Total possible score ranges between 0-100, with higher scores indicative of better outcomes.
Quality of Life After Brain Injury (QOLIBRI) | 3-months post-intervention
  Assesses quality of life. Total possible score ranges between 0-100, with higher scores indicative of better outcomes.
Headache Impact Test (HIT-6) | Baseline
  Assesses headache intensity. Total possible score ranges from 36-78, with higher scores indicative of worse outcomes.
Headache Impact Test (HIT-6) | Within 1 week post-intervention
  Assesses headache intensity. Total possible score ranges from 36-78, with higher scores indicative of worse outcomes.
Headache Impact Test (HIT-6) | 1-month post-intervention
  Assesses headache intensity. Total possible score ranges from 36-78, with higher scores indicative of worse outcomes.
Headache Impact Test (HIT-6) | 3-months post-intervention
  Assesses headache intensity. Total possible score ranges from 36-78, with higher scores indicative of worse outcomes.
Patient Health Questionnaire (PHQ-9) | Baseline
  Assesses depressive symptoms. Total possible score ranges from 0-27, with higher scores indicative of worse outcomes.
Patient Health Questionnaire (PHQ-9) | Within 1 week post-intervention
  Assesses depressive symptoms. Total possible score ranges from 0-27, with higher scores indicative of worse outcomes.
Patient Health Questionnaire (PHQ-9) | 1-month post-intervention
  Assesses depressive symptoms. Total possible score ranges from 0-27, with higher scores indicative of worse outcomes.
Patient Health Questionnaire (PHQ-9) | 3-months post-intervention
  Assesses depressive symptoms. Total possible score ranges from 0-27, with higher scores indicative of worse outcomes.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline
  Assesses feelings of anxiety. Total possible score ranges from 0-21, with higher scores indicative of worse outcomes.
Generalized Anxiety Disorder-7 (GAD-7) | Within 1 week post-intervention
  Assesses feelings of anxiety. Total possible score ranges from 0-21, with higher scores indicative of worse outcomes.
Generalized Anxiety Disorder-7 (GAD-7) | 1-month post-intervention
  Assesses feelings of anxiety. Total possible score ranges from 0-21, with higher scores indicative of worse outcomes.
Generalized Anxiety Disorder-7 (GAD-7) | 3-months post-intervention
  Assesses feelings of anxiety. Total possible score ranges from 0-21, with higher scores indicative of worse outcomes.
Screening for Somatoform Symptoms-7 (SOMS-7 CD Sub-scale) | Baseline
  Evaluates somatic symptoms. Total possible score ranges from 0-56, with higher scores indicative of worse outcomes.
Screening for Somatoform Symptoms-7 (SOMS-7 CD Sub-scale) | Within 1 week post-intervention
  Evaluates somatic symptoms. Total possible score ranges from 0-56, with higher scores indicative of worse outcomes.
Screening for Somatoform Symptoms-7 (SOMS-7 CD Sub-scale) | 1-month post-intervention
  Evaluates somatic symptoms. Total possible score ranges from 0-56, with higher scores indicative of worse outcomes.
Screening for Somatoform Symptoms-7 (SOMS-7 CD Sub-scale) | 3-months post-intervention
  Evaluates somatic symptoms. Total possible score ranges from 0-56, with higher scores indicative of worse outcomes.
Saint Louis University Mental Status Examination (SLUMS) | Baseline
  Assesses for mild cognitive impairment. Total possible score ranges from 0 to 30, with higher scores indicative of better outcomes.
Saint Louis University Mental Status Examination (SLUMS) | Within 1 week post-intervention
  Assesses for mild cognitive impairment. Total possible score ranges from 0 to 30, with higher scores indicative of better outcomes.
Saint Louis University Mental Status Examination (SLUMS) | 1-month post-intervention
  Assesses for mild cognitive impairment. Total possible score ranges from 0 to 30, with higher scores indicative of better outcomes.
Saint Louis University Mental Status Examination (SLUMS) | 3-months post-intervention
  Assesses for mild cognitive impairment. Total possible score ranges from 0 to 30, with higher scores indicative of better outcomes.
British Columbia Post-concussion Symptom Inventory | Baseline
  Assesses the frequency and intensity of post-concussion symptoms. Total possible score ranges from 3-67, with higher scores indicative of worse outcomes.
British Columbia Post-concussion Symptom Inventory | Within 1 week post-intervention
  Assesses the frequency and intensity of post-concussion symptoms. Total possible score ranges from 3-67, with higher scores indicative of worse outcomes.
British Columbia Post-concussion Symptom Inventory | 1-month post-intervention
  Assesses the frequency and intensity of post-concussion symptoms. Total possible score ranges from 3-67, with higher scores indicative of worse outcomes.
British Columbia Post-concussion Symptom Inventory | 3-months post-intervention
  Assesses the frequency and intensity of post-concussion symptoms. Total possible score ranges from 3-67, with higher scores indicative of worse outcomes.
Post-traumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Baseline
  Assesses PTSD symptoms. Total possible score ranges from 0-80, with higher scores indicative of worse outcomes.
Post-traumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Within 1 week post-intervention
  Assesses PTSD symptoms. Total possible score ranges from 0-80, with higher scores indicative of worse outcomes.
Post-traumatic Stress Disorder Checklist for DSM-5 (PCL-5) | 1-month post-intervention
  Assesses PTSD symptoms. Total possible score ranges from 0-80, with higher scores indicative of worse outcomes.
Post-traumatic Stress Disorder Checklist for DSM-5 (PCL-5) | 3-months post-intervention
  Assesses PTSD symptoms. Total possible score ranges from 0-80, with higher scores indicative of worse outcomes.
Patient Health Questionnaire-15 (PHQ-15) | Baseline
  Assesses somatic symptoms. Total possible score ranges from 0-30, with higher scores indicative of worse outcomes.
Patient Health Questionnaire-15 (PHQ-15) | Within 1 week post-intervention
  Assesses somatic symptoms. Total possible score ranges from 0-30, with higher scores indicative of worse outcomes.
Patient Health Questionnaire-15 (PHQ-15) | 1-month post-intervention
  Assesses somatic symptoms. Total possible score ranges from 0-30, with higher scores indicative of worse outcomes.
Patient Health Questionnaire-15 (PHQ-15) | 3-months post-intervention
  Assesses somatic symptoms. Total possible score ranges from 0-30, with higher scores indicative of worse outcomes.
Sleep and Concussion Questionnaire | Baseline
  Assesses sleep changes following mTBI. Total possible score ranges from 0-36, with higher scores indicative of worse outcomes.
Sleep and Concussion Questionnaire | Within 1 week post-intervention
  Assesses sleep changes following mTBI. Total possible score ranges from 0-36, with higher scores indicative of worse outcomes.
Sleep and Concussion Questionnaire | 1-month post-intervention
  Assesses sleep changes following mTBI. Total possible score ranges from 0-36, with higher scores indicative of worse outcomes.
Sleep and Concussion Questionnaire | 3-months post-intervention
  Assesses sleep changes following mTBI. Total possible score ranges from 0-36, with higher scores indicative of worse outcomes.
Brief Trauma Questionnaire | Baseline
  Assesses trauma history in a YES/NO format.
Brief Trauma Questionnaire | Within 1 week post-intervention
  Assesses trauma history in a YES/NO format.
Brief Trauma Questionnaire | 1-month post-intervention
  Assesses trauma history in a YES/NO format.
Brief Trauma Questionnaire | 3-months post-intervention
  Assesses trauma history in a YES/NO format.
Life Stress Questionnaire | Baseline
  Assesses significant life stressors in the past 2 years. Total possible score ranges from 0-1645, with higher scores indicative of worse outcomes.
Life Stress Questionnaire | Within 1 week post-intervention
  Assesses significant life stressors in the past 2 years. Total possible score ranges from 0-1645, with higher scores indicative of worse outcomes.
Life Stress Questionnaire | 1-month post-intervention
  Assesses significant life stressors in the past 2 years. Total possible score ranges from 0-1645, with higher scores indicative of worse outcomes.
Life Stress Questionnaire | 3-months post-intervention
  Assesses significant life stressors in the past 2 years. Total possible score ranges from 0-1645, with higher scores indicative of worse outcomes.
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline
  Assesses PTSD symptoms over the past week. Total possible symptom severity score ranges from 0-80, with higher scores indicative of worse outcomes.
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Within 1 week post-intervention
  Assesses PTSD symptoms over the past week. Total possible symptom severity score ranges from 0-80 with higher scores indicative of worse outcomes.
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | 1-month post-intervention
  Assesses PTSD symptoms over the past week. Total possible symptom severity score ranges from 0-80 with higher scores indicative of worse outcomes.
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | 3-months post-intervention
  Assesses PTSD symptoms over the past week. Total possible symptom severity score ranges from 0-80 with higher scores indicative of worse outcomes.
Montgomery-Asberg Depression Rating Scale | Baseline
  Semi-structured interview to assess depression symptoms. Total possible score ranges from 0-60, with higher scores indicative of worse outcomes.
Montgomery-Asberg Depression Rating Scale | Within 1 week post-intervention
  Semi-structured interview to assess depression symptoms. Total possible score ranges from 0-60, with higher scores indicative of worse outcomes.
Montgomery-Asberg Depression Rating Scale | 1-month post-intervention
  Semi-structured interview to assess depression symptoms. Total possible score ranges from 0-60, with higher scores indicative of worse outcomes.
Montgomery-Asberg Depression Rating Scale | 3-months post-intervention
  Semi-structured interview to assess depression symptoms. Total possible score ranges from 0-60, with higher scores indicative of worse outcomes.
Columbia Suicide Severity Rating Scale | Baseline
  Screening tool for suicidal ideation and behavior
Columbia Suicide Severity Rating Scale | Within 1 week post-intervention
  Screening tool for suicidal ideation and behavior
Columbia Suicide Severity Rating Scale | 1-month post-intervention
  Screening tool for suicidal ideation and behavior
Columbia Suicide Severity Rating Scale | 3-months post-intervention
  Screening tool for suicidal ideation and behavior

OTHER OUTCOMES:
Functional near infrared spectroscopy | Baseline
  Functional near infrared spectroscopy (fNIRS) will used as a tool to determine TMS response
Functional near infrared spectroscopy | Within 1 week post-intervention
  Functional near infrared spectroscopy (fNIRS) will used as a tool to determine TMS response
Functional near infrared spectroscopy | 1-month post-intervention
  Functional near infrared spectroscopy (fNIRS) will used as a tool to determine TMS response
Functional near infrared spectroscopy | 3-months post-intervention
  Functional near infrared spectroscopy (fNIRS) will used as a tool to determine TMS response

CONTACTS AND LOCATIONS:
Overall Officials: Chantel T Debert, MD MSc FRCPC CSCN, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maas AIR, Menon DK, Adelson PD, Andelic N, Bell MJ, Belli A, Bragge P, Brazinova A, Buki A, Chesnut RM, Citerio G, Coburn M, Cooper DJ, Crowder AT, Czeiter E, Czosnyka M, Diaz-Arrastia R, Dreier JP, Duhaime AC, Ercole A, van Essen TA, Feigin VL, Gao G, Giacino J, Gonzalez-Lara LE, Gruen RL, Gupta D, Hartings JA, Hill S, Jiang JY, Ketharanathan N, Kompanje EJO, Lanyon L, Laureys S, Lecky F, Levin H, Lingsma HF, Maegele M, Majdan M, Manley G, Marsteller J, Mascia L, McFadyen C, Mondello S, Newcombe V, Palotie A, Parizel PM, Peul W, Piercy J, Polinder S, Puybasset L, Rasmussen TE, Rossaint R, Smielewski P, Soderberg J, Stanworth SJ, Stein MB, von Steinbuchel N, Stewart W, Steyerberg EW, Stocchetti N, Synnot A, Te Ao B, Tenovuo O, Theadom A, Tibboel D, Videtta W, Wang KKW, Williams WH, Wilson L, Yaffe K; InTBIR Participants and Investigators. Traumatic brain injury: integrated approaches to improve prevention, clinical care, and research. Lancet Neurol. 2017 Dec;16(12):987-1048. doi: 10.1016/S1474-4422(17)30371-X. Epub 2017 Nov 6. No abstract available. PMID 29122524
- [Background] Hunt C, Zanetti K, Kirkham B, Michalak A, Masanic C, Vaidyanath C, Bhalerao S, Cusimano MD, Baker A, Ouchterlony D. Identification of hidden health utilization services and costs in adults awaiting tertiary care following mild traumatic brain injury in Toronto, Ontario, Canada. Concussion. 2016 Aug 8;1(4):CNC21. doi: 10.2217/cnc-2016-0009. eCollection 2016 Dec. PMID 30202563
- [Background] Hendrikse J, Kandola A, Coxon J, Rogasch N, Yucel M. Combining aerobic exercise and repetitive transcranial magnetic stimulation to improve brain function in health and disease. Neurosci Biobehav Rev. 2017 Dec;83:11-20. doi: 10.1016/j.neubiorev.2017.09.023. Epub 2017 Sep 23. PMID 28951250
- [Background] Daoud H, Alharfi I, Alhelali I, Charyk Stewart T, Qasem H, Fraser DD. Brain injury biomarkers as outcome predictors in pediatric severe traumatic brain injury. Neurocrit Care. 2014 Jun;20(3):427-35. doi: 10.1007/s12028-013-9879-1. PMID 23943317
- [Background] Mychasiuk R, Hehar H, Ma I, Kolb B, Esser MJ. The development of lasting impairments: a mild pediatric brain injury alters gene expression, dendritic morphology, and synaptic connectivity in the prefrontal cortex of rats. Neuroscience. 2015 Mar 12;288:145-55. doi: 10.1016/j.neuroscience.2014.12.034. Epub 2014 Dec 30. PMID 25555930
- [Background] Henry LC, Tremblay S, Boulanger Y, Ellemberg D, Lassonde M. Neurometabolic changes in the acute phase after sports concussions correlate with symptom severity. J Neurotrauma. 2010 Jan;27(1):65-76. doi: 10.1089/neu.2009.0962. PMID 19761385
- [Background] Liu G, Feng D, Wang J, Zhang H, Peng Z, Cai M, Yang J, Zhang R, Wang H, Wu S, Tan Q. rTMS Ameliorates PTSD Symptoms in Rats by Enhancing Glutamate Transmission and Synaptic Plasticity in the ACC via the PTEN/Akt Signalling Pathway. Mol Neurobiol. 2018 May;55(5):3946-3958. doi: 10.1007/s12035-017-0602-7. Epub 2017 May 26. PMID 28550530
- [Background] Lewis CP, Port JD, Frye MA, Vande Voort JL, Ameis SH, Husain MM, Daskalakis ZJ, Croarkin PE. An Exploratory Study of Spectroscopic Glutamatergic Correlates of Cortical Excitability in Depressed Adolescents. Front Neural Circuits. 2016 Nov 29;10:98. doi: 10.3389/fncir.2016.00098. eCollection 2016. PMID 27965544
- [Background] Yang XR, Kirton A, Wilkes TC, Pradhan S, Liu I, Jaworska N, Damji O, Keess J, Langevin LM, Rajapakse T, Lebel RM, Sembo M, Fife M, MacMaster FP. Glutamate alterations associated with transcranial magnetic stimulation in youth depression: a case series. J ECT. 2014 Sep;30(3):242-7. doi: 10.1097/YCT.0000000000000094. PMID 24820947
- [Background] Covassin T, Elbin RJ 3rd, Larson E, Kontos AP. Sex and age differences in depression and baseline sport-related concussion neurocognitive performance and symptoms. Clin J Sport Med. 2012 Mar;22(2):98-104. doi: 10.1097/JSM.0b013e31823403d2. PMID 22246342
- [Background] Harmon KG, Drezner JA, Gammons M, Guskiewicz KM, Halstead M, Herring SA, Kutcher JS, Pana A, Putukian M, Roberts WO. American Medical Society for Sports Medicine position statement: concussion in sport. Br J Sports Med. 2013 Jan;47(1):15-26. doi: 10.1136/bjsports-2012-091941. PMID 23243113
- [Background] McCrory P, Meeuwisse WH, Aubry M, Cantu RC, Dvorak J, Echemendia RJ, Engebretsen L, Johnston KM, Kutcher JS, Raftery M, Sills A, Benson BW, Davis GA, Ellenbogen R, Guskiewicz KM, Herring SA, Iverson GL, Jordan BD, Kissick J, McCrea M, McIntosh AS, Maddocks DL, Makdissi M, Purcell L, Putukian M, Schneider K, Tator CH, Turner M. Consensus statement on concussion in sport--the 4th International Conference on Concussion in Sport held in Zurich, November 2012. PM R. 2013 Apr;5(4):255-79. doi: 10.1016/j.pmrj.2013.02.012. Epub 2013 Feb 27. No abstract available. PMID 23466418
- [Background] Covassin T, Elbin RJ, Harris W, Parker T, Kontos A. The role of age and sex in symptoms, neurocognitive performance, and postural stability in athletes after concussion. Am J Sports Med. 2012 Jun;40(6):1303-12. doi: 10.1177/0363546512444554. Epub 2012 Apr 26. PMID 22539534
- [Background] Scholkmann F, Kleiser S, Metz AJ, Zimmermann R, Mata Pavia J, Wolf U, Wolf M. A review on continuous wave functional near-infrared spectroscopy and imaging instrumentation and methodology. Neuroimage. 2014 Jan 15;85 Pt 1:6-27. doi: 10.1016/j.neuroimage.2013.05.004. Epub 2013 May 16. PMID 23684868
- [Background] Kleinschmidt A, Obrig H, Requardt M, Merboldt KD, Dirnagl U, Villringer A, Frahm J. Simultaneous recording of cerebral blood oxygenation changes during human brain activation by magnetic resonance imaging and near-infrared spectroscopy. J Cereb Blood Flow Metab. 1996 Sep;16(5):817-26. doi: 10.1097/00004647-199609000-00006. PMID 8784226
- [Background] Hocke LM, Duszynski CC, Debert CT, Dleikan D, Dunn JF. Reduced Functional Connectivity in Adults with Persistent Post-Concussion Symptoms: A Functional Near-Infrared Spectroscopy Study. J Neurotrauma. 2018 Jun 1;35(11):1224-1232. doi: 10.1089/neu.2017.5365. Epub 2018 Mar 23. PMID 29373947
- [Background] Santosa H, Fishburn F, Zhai X, Huppert TJ. Investigation of the sensitivity-specificity of canonical- and deconvolution-based linear models in evoked functional near-infrared spectroscopy. Neurophotonics. 2019 Apr;6(2):025009. doi: 10.1117/1.NPh.6.2.025009. Epub 2019 May 30. PMID 31172019
- [Background] Huppert TJ, Diamond SG, Franceschini MA, Boas DA. HomER: a review of time-series analysis methods for near-infrared spectroscopy of the brain. Appl Opt. 2009 Apr 1;48(10):D280-98. doi: 10.1364/ao.48.00d280. PMID 19340120
- [Background] Kontos AP, Huppert TJ, Beluk NH, Elbin RJ, Henry LC, French J, Dakan SM, Collins MW. Brain activation during neurocognitive testing using functional near-infrared spectroscopy in patients following concussion compared to healthy controls. Brain Imaging Behav. 2014 Dec;8(4):621-34. doi: 10.1007/s11682-014-9289-9. PMID 24477579
- [Background] Wu Z, Mazzola CA, Catania L, Owoeye O, Yaramothu C, Alvarez T, Gao Y, Li X. Altered cortical activation and connectivity patterns for visual attention processing in young adults post-traumatic brain injury: A functional near infrared spectroscopy study. CNS Neurosci Ther. 2018 Jun;24(6):539-548. doi: 10.1111/cns.12811. Epub 2018 Jan 22. PMID 29359534
- [Derived] du Plessis S, Oni IK, Lapointe AP, Campbell C, Dunn JF, Debert CT. Treatment of Persistent Postconcussion Syndrome With Repetitive Transcranial Magnetic Stimulation Using Functional Near-Infrared Spectroscopy as a Biomarker of Response: Protocol for a Randomized Controlled Clinical Trial. JMIR Res Protoc. 2022 Mar 22;11(3):e31308. doi: 10.2196/31308. PMID 35315783